CLINICAL TRIAL: NCT05558917
Title: Comparison Between PECS BLOCK 2 vs ESP BLOCK in Ocnologic Breast Surgery: Randomized Controlled Trial on Postoperatory Oppioid Consumption
Brief Title: Comparison Between PECS BLOCK 2 vs ESP BLOCK in Ocnologic Breast Surgery
Acronym: ESPECS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ASO.RianGen.22.02
Record Dates: First submitted 2022-09-07; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Carcinoma
Keywords: PECS2; ESP BLOCK; Breast Anesthesia; Mastectomy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS BLOCK 2 (Active Comparator): PECS 2 (or modified PECS) is a block that involves the administration of local anesthetic under ultrasound guidance between the great pectoral and small pectoral and between the small pectoral and serratus anterior.
  Interventions: Procedure: PECS BLOCK 2
- ESP BLOCK (Experimental): ESP block is a block that involves injection of local anesthetic below the elevator muscles of the spine.
  Interventions: Procedure: ESP BLOCK

INTERVENTIONS:
Procedure: PECS BLOCK 2 — With the patient supine, the linear probe will be placed in the sagittal plane slightly lateral to the hemiclavicular line ipsilateral to the surgical site. Once both muscle planes of interest have been identified, in-plane needle insertion will proceed in the cranio-caudal direction. The first local anesthetic administration with Ropivacaine 0.5% will be 20ml between small pectoralis and serratus anterior. Coming out with the needle, 10ml of Ropivacaine 0.5% will then be injected between large and small pectoral.
  Arms: PECS BLOCK 2
Procedure: ESP BLOCK — Positioning yourself behind the patient, lying on her side with the surgical hemilateral on top, you place the linear ultrasound probe in the sagittal plane and find the lateral margin of the transverse process. At this point, the blocking needle is inserted in the caudocranial direction and 25ml of Ropivacaine 0.5% is injected, taking care to visualize the anesthetic spread in the cranial direction.
  Arms: ESP BLOCK

SUMMARY:
The study aims to compare the efficacy of the two operating blocks PECS2 and ESP by measuring postoperative opioid consumption and, secondarily, to compare (between PECS and ESP) postoperative opioid consumption between surgery with/without axillary cavity dissection and with/without implantation of prosthesis or expansion

DETAILED DESCRIPTION:
Breast cancer is the most frequent type of cancer in the female population. Early detection is the most effective tool for improving prognosis, and the surgical approach plays a central role in the treatment of this disease. However, many are the psychophysical implications that patients face: among the main ones is postoperative and chronic pain, a symptom that greatly worsens the quality of life.

In the last decade it has been witnessed an important development of locoregional anesthesia techniques in all surgeries. In breast surgery, particularly mastectomy, the following locoregional anesthesia techniques are referred to as the Gold Standard:

1. PVB (Paravertebral Block)
2. PECS2 BLOCK (or modified PECS). For the same purposes, ESP Block (Erector Spinae Plane Block) has been applied experimentally, which has already shown its effectiveness in breast surgery in several trials.

By comparing postoperative opioid consumption between the two groups of patients, divided into PECS Block and ESP Block, the study aims to identify which anesthesia block is most effective in order to improve the care of patients undergoing mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mastectomy exclusively for breast cancer
* Presence of written informed consent to the trial

Exclusion Criteria:

* Bilateral breast surgery
* Previous drug use
* Chronic opioid and minor opioid therapy
* BMI >40
* Allergy or contraindications to taking Paracetamol and Toradol
* Inability to use PCA (Patient Controlled Analgesia)
* Intraoperative opioid administration
* Patients with neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-09-07 (Estimated); Study Completion 2023-11-07 (Estimated)

PRIMARY OUTCOMES:
Morphine equivalent consumption in the postoperative 24h in simple mastectomies | Postoperative 24 hours
  Morphine-equivalent consumption in the postoperative 24h that patients self-administer between the group of patients undergoing ESP and those undergoing PECS 2 in simple mastectomies.

SECONDARY OUTCOMES:
Morphine-equivalent consumption in the postoperative 24h in mastectomies with axillary cavity emptying | Postoperative 24 hours
  Morphine-equivalent consumption in the postoperative 24h that patients self-administer between the group of patients undergoing ESP and those undergoing PECS 2 in mastectomies with axillary cavity emptying.
Morphine-equivalent consumption in the postoperative 24h in mastectomies with prosthesis or expander placement | Postoperative 24 hours
  Consumption of morphine equivalents in the postoperative 24h that patients self-administer between the group of patients undergoing ESP and those undergoing PECS 2 in astecctomies with prosthesis or expander placement.
Morphine-equivalent consumption in the postoperative 24h in mastectomies with axillary cavity emptying and implantation of prosthesis or expander | Postoperative 24 hours
  Consumption of morphine equivalents in the postoperative 24h that patients self-administer between the group of patients undergoing ESP and those undergoing PECS 2 in mastectomies with axillary cavity emptying and implantation of prosthesis or expander
PONV (Post Operating Nausea and Vomiting) | Immediately after the surgery and at 2-4-8-12-24 hours after surgery
  Number of times the patient experienced nausea or vomiting
Complications incidence | Postoperative 24 hours
  Number of times the patient experienced complications such as bleeding or pneumothorax
Time from end of surgery to first walk | Postoperative 72 hours
  Time in hours
Length of hospitalization | Up to 7 days
  Lenght in days
Patient's Likert Scale | Postoperative 24 hours
  Patient satisfaction, from 1 - Strongly disagree to 5 - Strongly agree
Surgeon's Likert scale | Postoperative 24 hours
  Surgeon satisfaction, from 1 - Strongly disagree to 5 - Strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Mirco Leo, Physician, Principal Investigator — Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo
Locations (1):
- Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont, Italy